CLINICAL TRIAL: NCT03886025
Title: The Use of Combined Anodal Transcranial Direct Current Stimulation (tDCS) and Cognitive Training to Modulate Decision-making in Healthy People
Brief Title: Combined Anodal Transcranial Direct Current Stimulation (tDCS) and Cognitive Training and Decision-making
Acronym: tDCS-CTDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Najat Khalifa (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor-Investigator, Dr. Najat Khalifa, Associate Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6025821
Record Dates: First submitted 2019-03-15; First posted 2019-03-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Impulsivity; Decision Making
Keywords: transcranial Direct Current Stimulation (tDCS); Decision-making; Implusivity; Brain stimulation
MeSH Terms: conditions — Impulsive Behavior | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Intervention Model Description: Single blind Randomized Controlled Trial
Who Masked: Participant
Masking Description: Participants will be randomly assigned to receive either combined anodal tDCS and cognitive training or combined sham tDCS and cognitive training. The participants will be blind to whether the tDCS is active or sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined anodal tDCS and cognitive training (Experimental): Combined anodal tDCS and cognitive training. Anodal tDCS will be delivered while the participant is completing the cognitive training task (Iowa Gambling Task). Anodal tDCS will use a constant current of 2mA, delivered via gradual increase and decrease over 10 seconds at the onset and offset of stimulation (current ramps), respectively. The duration of each tDCS session will be 20 minutes.
  Interventions: Other: Anodal transcranial Direct Current Stimulation (tDCS); Behavioral: Cognitive training
- Combined sham tDCS and cognitive training (Sham Comparator): Combined sham tDCS and cognitive training. Sham tDCS will be delivered while the participant is completing the cognitive training task (Iowa Gambling Task). For sham tDCS, the current will be delivered only in the first 10 seconds, after which the stimulation will cease but with the electrodes still in place throughout the session. The duration of each tDCS session will be 20 minutes.
  Interventions: Behavioral: Cognitive training; Other: Sham transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Other: Anodal transcranial Direct Current Stimulation (tDCS) — Non-invasive brain stimulation
  Arms: Combined anodal tDCS and cognitive training
Behavioral: Cognitive training — Iowa Gambling Task will be used for cognitive training
Other: Sham transcranial Direct Current Stimulation (tDCS) — Non-invasive brain stimulation
  Arms: Combined sham tDCS and cognitive training

SUMMARY:
This study aims to (i) assess the effects of combined tDCS and cognitive training on decision-making on a trained task (Iowa Gambling Task; IGT); and (ii) test generalization to a closely related cognitive domain, namely motor impulsivity. It is hypothesized that combined anodal tDCS and cognitive training will result in more advantageous decisions and better impulse control than combined sham tDCS and cognitive training.

DETAILED DESCRIPTION:
Impaired decision-making under conditions of uncertainty and risk has been implicated in maladaptive personality development and violent behaviour. There is a dearth of studies that examined the effects of combined tDCS and cognitive training on decision-making under conditions of uncertainty and risk. It is also unclear if these effects are generalizable to tasks in other domains such as response inhibition (motor impulsivity).

To examine these issues further, a single blind parallel arms randomized controlled trial will be conducted, involving a sample of healthy volunteers aged between 18 and 40. This will entail applying either active or sham tDCS over the anterior frontal cortex (including the vm-PFC) while participants undertake decision-making training using the Iowa Gambling Task. Decision-making will be assessed using the IGT, which is a computerized gambling task used to assess decision-making under conditions of uncertainty and risk. IGT is sensitive to damage to the ventromedial prefrontal cortex (vmPFC), which is considered to play a key role in decision-making. Motor impulsivity will be measured using the Stop Signal Task (SST). The UPPS+P Impulsive Behaviour Scale will be used to index trait impulsivity. The Profile of Mood States will be used to measure state emotion before and after tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Consenting volunteers aged between 18 and 40.

Exclusion Criteria:

* Individuals with epilepsy, other neurological conditions and history of significant head injury will be excluded.
* Individuals with a history of substance misuse, major mental disorder and those receiving psychotropic medication will be also excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Iowa Gambling Task (IGT) net scores | Change from baseline after 20 minutes of combined cognitive training and tDCS stimulation
  IGT is a measure of decision making under conditions of uncertainty and risk.

SECONDARY OUTCOMES:
Stop Signal Task (SST) reaction time | Change from baseline after 20 minutes of combined cognitive training and tDCS stimulation
  SST is a measure of inhibitory control
Urgency, Perseveration, Premeditation, Sensation Seeking + Positive Urgency (UPPS+P) Impulsive Behavior Scale total scores | Baseline
  UPPS+P is a 59 item self-report measure of trait impulsivity. Each item is rated on a scale of 1-4 (1= totally disagree, 4=totally agree) yielding a total score out of 216 (range=59 - 216) Higher scores denote higher impulsivity.
Abbreviated Profile of Mood States (POMS) Total Mood Disturbance score | Baseline
  Abbreviated POMS is a 40-item measure of current mood states. Each item is rated on a scale of 0-4 (0=Not at all, 4=Extremely). The total Mood Disturbance score is calculated by summing the totals for the negative subscales (tension, depression, anger, fatigue, confusion) and then subtracting the totals for the positive subscales (vigour, esteem related affect) and then adding a constant 100. Higher scores denote greater mood disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Najat Khalifa, MD, Principal Investigator — Queen's University - Canada
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared with researchers other than the study investigators.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03886025/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03886025/ICF_001.pdf